CLINICAL TRIAL: NCT00671255
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Outpatient, Safety and Efficacy Study of TAK-375 in Elderly Subjects With Chronic Insomnia
Brief Title: Safety and Efficacy of Ramelteon in Elderly Subjects With Chronic Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-02-TL-375-025; U1111-1114-1190 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Insomnia
Keywords: Chronic Insomnia; Drug Therapy; Elderly
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ramelteon 4 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 4 mg, tablets, orally, once daily for up to 5 weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 4 mg QD
Drug: Ramelteon — Ramelteon 8 mg, tablets, orally, once daily for up to 5 weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 8 mg QD
Drug: Placebo — Ramelteon placebo-matching, tablets, orally, each night for up to 35 consecutive days.
  Arms: Placebo

SUMMARY:
This purpose of this study is to evaluate the safety and effectiveness of Ramelteon, once daily (QD), in elderly participants with chronic insomnia.

DETAILED DESCRIPTION:
Insomnia is characterized by a complaint of initiating and maintaining sleep or complaints of nonrestorative and non-refreshing sleep. Transient insomnia affects approximately one-third to one-half of the US population, based on the results of 2 surveys of representative samples of the adult US population conducted by the Gallup Organization in which respondents were asked if they had "ever had difficulty sleeping." Based on reports of "regular" or "frequent" sleep difficulty, results from the same studies suggest that approximately one-tenth of the US population experiences chronic insomnia. The ideal treatment for insomnia would reduce the latency to onset of sleep and increase total sleep time, without a negative impact on sleep architecture and without safety concerns or next-day effects.

Ramelteon is a selective melatonin-1 receptor agonist under development by Takeda Chemical Industries, Ltd., for the treatment of transient and chronic insomnia and for the treatment of Circadian Rhythm Sleep Disorders.

Ramelteon is the first candidate in a novel class of drugs based on this mechanism. Based on non-clinical and clinical studies completed to date, TAK-375 has the potential to offer unique advantages relative to approved hypnotics in terms of its pharmacological profile and its selectivity to the melatonin-1 receptor.

This study is designed to determine the safety and efficacy of 35-day treatment of chronic insomnia with ramelteon. Participation in this study is anticipated to be approximately 2 months.

ELIGIBILITY:
Inclusion Criteria

* Subject is a male or a post-menopausal female.
* Primary insomnia as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised for at least 3 months and a history of daytime complaint(s) associated with disturbed sleep.
* Subjective sleep latency greater than or equal to 45 minutes and a subjective total sleep time less than or equal to 6.5 hours per night for at least 3 nights during the week of the lead-in period.
* Habitual bedtime is between 8:30 PM and 12:00 AM.
* Body mass index between 18 and 34, inclusive.

Exclusion Criteria

* Known hypersensitivity to ramelteon or related compounds, including melatonin.
* Previously participated in a study involving ramelteon.
* Participated in any other investigational study, and/or took any investigational drug within 30 days or five half-lives prior to the first day of single-blind study medication, whichever is longer.
* Sleep schedule changes required by employment (eg, shift worker) within three months prior to the first day of single-blind study medication, or has flown across greater than three time zones within seven days prior to screening.
* Participated in a weight loss program or substantially altered exercise routine within 30 days prior to the first day of single blind study medication.
* Has ever had a history of seizures, sleep apnea, chronic obstructive pulmonary disease, restless leg syndrome, schizophrenia, bipolar disorder, mental retardation, or cognitive disorder.
* History of psychiatric disorder within the past 12 months.
* History of drug addiction or drug abuse within the past 12 months.
* History of alcohol abuse within the past 12 months, as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised and/or regularly consumes 4 or more alcoholic drinks per day.
* Current significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic or metabolic disease, unless currently controlled and stable with protocol-allowed medication.
* Uses tobacco products during nightly awakenings.
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Positive hepatitis panel.
* Any additional condition(s) that in the Investigator's opinion would:

  * affect sleep-wake function
  * prohibit the subject from completing the study
  * not be in the best interest of the subject.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication, including:

  * Anxiolytics
  * Hypnotics
  * Antidepressants
  * Anticonvulsants
  * Sedating H1 antihistamines
  * Systemic steroids
  * Respiratory stimulants
  * Decongestants
  * Over-the-counter and prescription stimulants
  * Over-the-counter and prescription diet aids
  * Central nervous system active drugs
  * Narcotic analgesics
  * All beta blockers
  * Melatonin
  * St. John's Wort
  * Kava-kava
  * Gingko biloba

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 829 (Actual)
Dates: Start 2002-12; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Mean Subjective Sleep Latency per subject diary, from Nights 1 through 7 of double-blind Treatment | Weeks 1, 2, 3, 4 and 5 or Final Visit.

SECONDARY OUTCOMES:
Subjective Total Sleep Time. | Weeks 1, 2, 3, 4 and 5 or Final Visit.
Subjective Number of Awakenings. | Weeks 1, 2, 3, 4 and 5 or Final Visit.
Subjective Ease of Falling Back to Sleep after Awakening. | Weeks 1, 2, 3, 4 and 5 or Final Visit.
Subjective Sleep Quality. | Weeks 1, 2, 3, 4 and 5 or Final Visit.
Clinical Global Impression Change of Condition. | Weeks 1, 2, 3, 4 and 5 or Final Visit.
Clinical Global Impression Severity of Illness. | Weeks 1, 2, 3, 4 and 5 or Final Visit.
Clinical Global Impression Therapeutic Effect. | Weeks 1, 2, 3, 4 and 5 or Final Visit.
Clinical Global Impression Side Effects. | Weeks 1, 2, 3, 4 and 5 or Final Visit.
Average Subjective Sleep Latency over the week preceding the Day 15, Day 22, Day 29, and Day 36 Visits. | Weeks 2, 3, 4 and 5 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (115):
- United States (102):
  - Columbiana, Alabama
  - Mobile, Alabama
  - Muscle Shoals, Alabama
  - Tallahassee, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tempe, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Encinitas, California
  - Irvine, California
  - La Jolla, California
  - La Mesa, California
  - Los Angeles, California
  - Murrieta, California
  - Northridge, California
  - Oakland, California
  - Redlands, California
  - Riverside, California
  - Rosemead, California
  - San Diego, California
  - Spring Valley, California
  - Vista, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Clearwater, Florida
  - DeLand, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Longwood, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Safety Harbor, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Blairsville, Georgia
  - Macon, Georgia
  - Chciago, Illinois
  - Northfield, Illinois
  - Evansville, Indiana
  - Shawnee Mission, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Murray, Kentucky
  - New Orleans, Louisiana
  - Bethesda, Maryland
  - Belmont, Massachusetts
  - Brockton, Massachusetts
  - Newton, Massachusetts
  - Detroit, Michigan
  - Hattiesburg, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Brick, New Jersey
  - Edison, New Jersey
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - Great Neck, New York
  - Manlius, New York
  - Mineola, New York
  - Williamsville, New York
  - Cary, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Beachwood, Ohio
  - Canfield, Ohio
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Jenkintown, Pennsylvania
  - Reading, Pennsylvania
  - Scotland, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Fayetteville, Tennessee
  - Johnson City, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Bellevue, Washington
  - Gig Harbor, Washington
  - Madison, Wisconsin
  - New Berlin, Wisconsin
- Canada (13):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Medicine Hat, Alberta
  - North Vancouver, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Corunna, Ontario
  - London, Ontario
  - North Bay, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Parkdale, Prince Edward Island
  - Montreal, Quebec

REFERENCES:
- [Result] Mini LJ, Wang-Weigand S, Zhang J. Self-reported efficacy and tolerability of ramelteon 8 mg in older adults experiencing severe sleep-onset difficulty. Am J Geriatr Pharmacother. 2007 Sep;5(3):177-84. doi: 10.1016/j.amjopharm.2007.09.004. PMID 17996657
- [Result] Roth T, Seiden D, Sainati S, Wang-Weigand S, Zhang J, Zee P. Effects of ramelteon on patient-reported sleep latency in older adults with chronic insomnia. Sleep Med. 2006 Jun;7(4):312-8. doi: 10.1016/j.sleep.2006.01.003. Epub 2006 May 18. PMID 16709464
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI